CLINICAL TRIAL: NCT02097277
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multiple Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamic Effects of BMS-986036 in Obese Adults With Type-2 Diabetes
Brief Title: A Study to Evaluate BMS-986036 in Obese Adults With Type-2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB130-002
Record Dates: First submitted 2014-03-19; First posted 2014-03-27 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pegbelfermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A: Placebo (Matching with BMS-986036 - Daily) (Placebo Comparator): Placebo (Matching with BMS-986036) 0 mg subcutaneous injection once daily for 12 weeks
  Interventions: Biological: Placebo (Matching with BMS-986036)
- Arm 2: Treatment B: BMS-986036 (1 mg Daily) (Experimental): BMS-986036 1 mg subcutaneous injection once daily for 12 weeks
  Interventions: Biological: BMS-986036
- Treatment C: BMS-986036 (5 mg Daily) (Experimental): BMS-986036 5 mg subcutaneous injection once daily for 12 weeks
  Interventions: Biological: BMS-986036
- Treatment D: BMS-986036 (20 mg Daily) (Experimental): BMS-986036 20 mg subcutaneous injection once daily for 12 weeks
  Interventions: Biological: BMS-986036
- Treatment E: BMS-986036 (20 mg Weekly) (Experimental): BMS-986036 20 mg subcutaneous injection once weekly (on Day 1 of each week) for 12 weeks
  Followed by Placebo (Matching with BMS-986036) 0 mg subcutaneous injection on Days 2-7 of each week for 12 weeks
  Interventions: Biological: BMS-986036; Biological: Placebo (Matching with BMS-986036)

INTERVENTIONS:
Biological: BMS-986036
  Arms: Arm 2: Treatment B: BMS-986036 (1 mg Daily); Treatment C: BMS-986036 (5 mg Daily); Treatment D: BMS-986036 (20 mg Daily); Treatment E: BMS-986036 (20 mg Weekly)
Biological: Placebo (Matching with BMS-986036)
  Arms: Treatment A: Placebo (Matching with BMS-986036 - Daily); Treatment E: BMS-986036 (20 mg Weekly)

SUMMARY:
The purpose of this study is to assess the potential of BMS-986036 for treatment obese adults with type-2 diabetes.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Diagnosed with type-2 diabetes mellitus with HbA1c ≥6.5% to less than 10.0%
* Body mass index 30.0 to 50.0

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Inability to self-administer subcutaneous injections
* Inability to be venipunctured
* Evidence of organ dysfunction beyond what is consistent with the target population
* History of allergy to PEGylated compounds or Fibroblast growth factor 21 (FGF21) related compounds

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2015-09-22 (Actual); Study Completion 2016-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- United States (9):
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Anaheim Clinical Trials Llc, Anaheim, California
  - National Research Institute, Los Angeles, California
  - Encompass Clinical Research, Spring Valley, California
  - All Medical Research, Llc, Cooper City, Florida
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Premier Research, Trenton, New Jersey
  - Metrolina Internal Medicine, Charlotte, North Carolina
  - Sterling Research Grp, Ltd., Cincinnati, Ohio
- Canada (6):
  - Manna Research Vancouver, Vancouver, British Columbia
  - Aggarwal And Associates, Brampton, Ontario
  - Rhodin Recherche Clinique, Drummondville, Quebec
  - Recherche Gcp Research, Montreal, Quebec
  - Alpha-Recherche Clinique, Québec, Quebec
  - Medexa Recherche, Victoriaville, Quebec

REFERENCES:
- [Derived] Charles ED, Neuschwander-Tetri BA, Pablo Frias J, Kundu S, Luo Y, Tirucherai GS, Christian R. Pegbelfermin (BMS-986036), PEGylated FGF21, in Patients with Obesity and Type 2 Diabetes: Results from a Randomized Phase 2 Study. Obesity (Silver Spring). 2019 Jan;27(1):41-49. doi: 10.1002/oby.22344. Epub 2018 Dec 6. PMID 30520566
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 219 participants were enrolled; 138 entered the lead-in period. Reasons for not entering lead-in period included "not meeting study eligibility criteria". 120 were randomized to treatment. Reasons not randomized: 6 withdrew consent, 2 lost to follow-up, 4 no longer met study criteria, 1 due to admin.reason by Sponsor and 4 due to other reasons.
Groups:
- Treatment A: Placebo: Placebo (Matching with BMS-986036) 0 mg subcutaneous injection once daily for 12 weeks.
- Treatment B: BMS-986036 (1 mg Daily): BMS-986036 1 mg subcutaneous injection once daily for 12 weeks.
Period: Overall Study
Arm/Group | Treatment A: Placebo | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Started | 24 | 24 | 24 | 24 | 24
Completed | 22 | 21 | 22 | 20 | 23
Not Completed | 2 | 3 | 2 | 4 | 1
Not completed — Subject no longer meets study criteria | 0 | 1 | 0 | 1 | 0
Not completed — Subject request to discontinue treatment | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A: Placebo | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly) | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (7.58) | 55.4 (9.44) | 55.3 (9.92) | 56.2 (8.17) | 55.2 (12.62) | 56.0 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 11 | 9 | 12 | 53
  Male | 14 | 13 | 13 | 15 | 12 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 2 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 3 | 2 | 5 | 15
  White | 22 | 20 | 18 | 20 | 15 | 95
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Glycosylated Hemoglobin A1c (HbA1c) From Baseline to Week 12
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Percent Change in Glycosylated Hemoglobin A1c (HbA1c) from Baseline to Week 12 was reported.
Time Frame: Baseline (Day 1) and Week 12
Population: The Pharmacodynamic Population included all subjects who received at least one dose of study medication and had PD biomarker data available, although only participants with both baseline and post-baseline data were included in the statistical analysis. Here, 'N' signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Treatment A: Placebo | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
Percent Change | 0.0005 (0.00622) | 0.0029 (0.00882) | 0.0007 (0.00692) | 0.0004 (0.00814) | -0.0004 (0.00418)

2. Secondary Outcome: Change in Body Weight From Baseline to Week 12
Description: Change in Body Weight from Baseline to Week 12 as a part of Physical measurement was reported.
Time Frame: Baseline (Day 1) and Week 12
Population: The Pharmacodynamic Population included all subjects who received at least one dose of study medication and had PD biomarker data available, although only subjects with both baseline and post-baseline data were included in the statistical analysis. Here, 'N' signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Treatment A: Placebo | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
Kilogram | -0.22 (2.615) | -0.26 (1.718) | -0.10 (2.883) | -1.09 (2.583) | -0.50 (2.297)

3. Secondary Outcome: Change From Baseline to Week 12 in Insulin Sensitivity Quantified by Composite Index of Insulin Sensitivity (CISI) (Matsuda Index)
Description: Whole body insulin sensitivity as quantified by Matsuda Index at the end of the treatment period, calculated by the following equation: 10,000/square root of(FPG*FI)*(FPG+PG30*2+PG60*3+PG120*2)/8*(FPI+PI30*2+PI60*3+PI120*2)/8). FPG=fasting plasma glucose level; FPI=fasting plasma insulin level; PG30,60,90, and 120=plasma glucose levels sampled at 30,60, and 120 minutes after oral glucose load; PI30,60,and 120=plasma insulin levels sampled at 30,60 and 120 minutes after the oral glucose load.
Time Frame: Baseline (Day 1) and Week 12
Population: The Pharmacodynamic Population included all participants who received at least one dose of study medication and had PD biomarker data available, although only participants with both baseline and post-baseline data were included in the statistical analysis. Here, 'N' signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Treatment A: Placebo | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
Unit on a scale | -0.18 (0.967) | -0.19 (1.348) | -0.18 (2.102) | 0.77 (2.455) | 0.54 (1.772)

4. Secondary Outcome: Change From Baseline to Week 12 in Insulin Sensitivity Quantified by Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: Homeostasis model assessment of insulin resistance (HOMA-IR) was used as a validated measure of insulin resistance. HOMA-IR is calculated using the following formula's fasting glucose(mg/dL) x fasting insulin(mU/L) / 405.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Unit on a Scale
Arm/Group | Treatment A: Placebo | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
Unit on a Scale | -0.19 (4.136) | 0.00 (5.633) | -1.88 (8.940) | -1.73 (4.589) | -0.34 (3.707)

5. Secondary Outcome: Change From Baseline to Week 12 in Insulin Sensitivity Quantified by Quantitative Insulin Sensitivity Check Index (QUICKI)
Description: The Quantitative Insulin Sensitivity Check Index (QUICKI) score, measures insulin sensitivity which is the inverse of insulin resistance. QUICKI is derived using the inverse of the sum of the logarithms of the fasting insulin and fasting glucose: 1 / (log(fasting insulin mU/L) + log(fasting glucose mg/dL)).
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Treatment A: Placebo | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
Unit on a scale | 0.00 (0.011) | 0.00 (0.010) | 0.00 (0.015) | 0.00 (0.016) | 0.00 (0.011)

6. Secondary Outcome: Change in Oral Glucose Tolerance Test (OGTT) Area Under the Curve From 0 to 2 Hours for Postprandial Glucose From Baseline to Week 12
Description: Blood samples were drawn after an overnight fast and standard OGTT from 0 to 120 minutes. Plasma Glucose levels over 2 hours were shown as Area Under the Curve, (AUC).
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimole*hour per Liter (mmol*hr/L)
Arm/Group | Treatment A: Placebo | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
Millimole*hour per Liter (mmol*hr/L) | 1.538 (4.2940) | 2.594 (5.8193) | -0.646 (7.0591) | -0.215 (4.7397) | -2.293 (4.9322)

7. Secondary Outcome: Change in OGTT Insulin AUC (0-2 Hours) From Baseline to Week 12
Description: Blood samples were drawn after an overnight fast and standard OGTT from 0 to 120 minutes. Insulin levels over 2 hours were shown as Area Under the Curve, (AUC).
Time Frame: Bseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol*hr/L
Arm/Group | Treatment A: Placebo | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
mmol*hr/L | -64.648 (231.6043) | -72.155 (277.4819) | -83.850 (215.3974) | -58.313 (205.1879) | -150.679 (257.5965)

8. Secondary Outcome: Change in OGTT C-peptide AUC (0-2 Hours) From Baseline to Week 12
Description: Blood samples were drawn after an overnight fast and standard OGTT from 0 to 120 minutes. C-peptide levels over 2 hours were shown as Area Under the Curve, (AUC).
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol*hr/L
Arm/Group | Treatment A: Placebo | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
mmol*hr/L | -0.287 (1.2463) | 0.031 (1.3926) | -0.181 (0.8927) | -0.169 (1.0176) | -0.750 (1.2224)

9. Secondary Outcome: Average Concentration (Cavg) of C-terminal Intact BMS-986036
Description: Cavg of C-terminal Intact BMS-986036 was reported.
Time Frame: Pre-dose, 6, 24 hours postdose on Week 8; pre-dose on Weeks 1, 2, 4, 6, 8, and 12; post treatment period on Week 13, 15 and 18 (Day 126)
Population: Serum concentration-time data will be used to develop a population PK model, and estimates of individual PK parameters will be derived from this model using a validated PK analysis program. Here, 'N' signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per Liter (ug/L)
Arm/Group | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 21 | 22 | 20 | 23
Microgram per Liter (ug/L) | 50.6 (60.6) | 204 (50.4) | 762 (49.2) | 197 (60.5)

10. Secondary Outcome: Maximum Observed Concentration (Cmax) of C-terminal Intact BMS-986036
Description: Maximum observed concentration (Cmax) of C-terminal Intact BMS-986036 was reported.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/liter
Arm/Group | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 21 | 22 | 20 | 23
microgram/liter | 53.3 (61.2) | 213 (50.4) | 807 (48.8) | 459 (41.4)

11. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours at Steady State (AUC [0-24 Hours, ss]) of C-terminal Intact BMS-986036
Description: AUC [0-24 hours, ss] of C-terminal Intact BMS-986036 was reported.
Time Frame: Pre-dose, 6, 24 hours postdose on Week 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/liter
Arm/Group | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 21 | 22 | 20 | 0
hour*microgram/liter | 1210 (60.6) | 4900 (50.4) | 18300 (49.2) |

12. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 168 Hours at Steady State (AUC [0-168 Hours, ss]) of C-terminal Intact BMS-986036
Description: AUC [0-168 hours, ss] of C-terminal Intact BMS-986036 was reported.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/liter
Arm/Group | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 0 | 0 | 0 | 23
hour*microgram/liter |  |  |  | 31800 (57.6)

13. Secondary Outcome: Average Concentration (Cavg) of Total BMS-986036
Description: Cavg of Total BMS-986036 was reported.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per Liter (ug/L)
Arm/Group | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 21 | 22 | 20 | 23
Microgram per Liter (ug/L) | 342 (42.3) | 1560 (44.6) | 6390 (43.2) | 1130 (38.9)

14. Secondary Outcome: Maximum Observed Concentration (Cmax) of Total BMS-986036
Description: Maximum observed concentration (Cmax) of Total BMS-986036 was reported.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/liter
Arm/Group | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 21 | 22 | 20 | 23
microgram/liter | 344 (42.5) | 1570 (44.5) | 6440 (43.1) | 1420 (36.1)

15. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours at Steady State (AUC [0-24 Hours, ss]) Total BMS-986036
Description: AUC [0-24 hours, ss] of Total BMS-986036 was reported.
Time Frame: Pre-dose, 6, 24 hours postdose on Week 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/liter
Arm/Group | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 21 | 22 | 20 | 0
hour*microgram/liter | 8200 (42.3) | 37400 (44.6) | 153000 (43.2) |

16. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 168 Hours at Steady State (AUC [0-168 Hours, ss]) of Total BMS-986036
Description: AUC [0-168 hours, ss] of Total BMS- 986036 was reported.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/liter
Arm/Group | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 0 | 0 | 0 | 23
hour*microgram/liter |  |  |  | 172000 (39.1)

17. Secondary Outcome: Percentage of Participants With ANTI-BMS-986036 Antibody Response
Description: Percentage of Participants with ANTI-BMS-986036 Antibody Response (ADA positive and ADA Negative) was reported. Participants were monitored for antibodies to BMS-986036 with an anti-BMS-986036 antibody assay. Titers were reported for samples testing positive in an assay.
Time Frame: Baseline and Day 126
Population: It included all treated participants who were randomized to treatment and subsequently received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
Number analyzed (Participants) | 24 | 24 | 24 | 24
Percentage of participants
  ADA Positive | 37.5 | 79.2 | 83.3 | 58.3
  ADA Negative | 62.5 | 16.7 | 12.5 | 37.5

ADVERSE EVENTS:
Time Frame: Approximately 2 years
Arm/Group | Treatment A: Placebo | Treatment B: BMS-986036 (1 mg Daily) | Treatment C: BMS-986036 (5 mg Daily) | Treatment D: BMS-986036 (20 mg Daily) | Treatment E: BMS-986036 (20 mg Weekly)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/24 | 0/24 | 1/24 | 0/24
Other Adverse Events (participants affected / at risk) | 9/24 | 12/24 | 7/24 | 10/24 | 10/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Placebo (N=24) | Treatment B: BMS-986036 (1 mg Daily) (N=24) | Treatment C: BMS-986036 (5 mg Daily) (N=24) | Treatment D: BMS-986036 (20 mg Daily) (N=24) | Treatment E: BMS-986036 (20 mg Weekly) (N=24)
Mitral Valve Disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tricuspid Valve Disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Placebo (N=24) | Treatment B: BMS-986036 (1 mg Daily) (N=24) | Treatment C: BMS-986036 (5 mg Daily) (N=24) | Treatment D: BMS-986036 (20 mg Daily) (N=24) | Treatment E: BMS-986036 (20 mg Weekly) (N=24)
Injection Site Bruising (General disorders) | 5 | 6 | 4 | 1 | 3
Injection Site Erythema (General disorders) | 1 | 1 | 0 | 2 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 2
Hunger (General disorders) | 0 | 0 | 2 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 1 | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 2 | 4 | 5
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 2 | 1 | 3 | 1 | 1
Headache (Nervous system disorders) | 2 | 1 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.